CLINICAL TRIAL: NCT01462552
Title: Assessment of Physician Compliance to Recommended Liver Function Test Monitoring for Tykerb Patients
Brief Title: Physician Liver Function Test (LFT) Monitoring for Tykerb Pts
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 115270; WEUKSTV4275 (Other: GSK); EPI40640 (Other: GSK)
Record Dates: First submitted 2011-05-19; First posted 2011-10-31 (Estimated); Last update posted 2015-04-15 (Estimated); Status verified 2015-04

CONDITIONS: Cancer
Keywords: liver function testing; Breast cancer; lapatanib
MeSH Terms: conditions — Neoplasms; Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Metastatic breast cancer pre-label group: Patients with metastatic breast cancer who initiated lapatanib between January 1, 2007 and December 31, 2007. Follow-up time for this group will continue until June 30, 2008 to allow these patients to have at least six months of follow-up time prior to the label change.
  Interventions: Drug: Lapatanib
- Metastatic breast cancer post-label group: Patients with metastatic breast cancer who initiated lapatanib between July 9, 2008 and December 31, 2009. Follow-up time for this group will continue until June 30, 2010 to allow these patients to have at least six month of follow-up.
  Interventions: Drug: Lapatanib

INTERVENTIONS:
Drug: Lapatanib — Prescription of lapatinib (Tykerb)

SUMMARY:
In July 2008, the lapatinib (Tykerb) Prescribing Information (label) was updated to include a boxed warning related to hepatotoxcity and detailed instructions for monitoring liver function before and during lapatanib exposure. For patient safety, it is of interest to know the extent to which providers are adherent with these guidelines for hepatic monitoring of lapatanib users.

Thus, the aim of this study is to determine if physicians conduct liver function testing prior to prescribing lapatanib and at regular intervals during exposure, and if they withdraw lapatanib, and do not re-treat, for patients who demonstrate severe liver enzyme elevations while exposed. These aims will be tested in the "Pre-label" (prior to the boxed warning) and "Post-label" (after the boxed warning) periods to determine if physician adherence to the guidelines changed as a result of the warning.

Specifically, the boxed warning provided the following guidance:

"Hepatotoxicity (alanine transaminase or aspartate transaminase >3 times the upper limit of normal and total bilirubin >1.5 times the upper limit of normal) has been observed in clinical trials (<1% of patients) and postmarketing experience. The hepatotoxicity may be severe and deaths have been reported. Causality of the deaths is uncertain. The hepatotoxicity may occur days to several months after initiation of treatment. Liver function tests (transaminases, bilirubin, and alkaline phosphatase) should be monitored before initiation of treatment, every 4 to 6 weeks during treatment, and as clinically indicated. If changes in liver function are severe, therapy with lapatanib should be discontinued and patients should not be re-treated with lapatanib"

The following objectives will be assessed and compared among patients prescribed lapatanib before and after the addition of detailed guidance on liver function testing to the product label on July 9, 2008:

1. Objective 1: Determine if physicians perform liver funtion tests (LFTs) prior to prescribing lapatanib (baseline)
2. Objective 2: Describe the prevalence of LFT elevations at baseline
3. Objective 3: Determine if physicians routinely perform LFTs during the duration of lapatanib exposure
4. Objective 4: Describe the cumulative incidence and incidence rate of LFT elevations during lapatanib exposure
5. Objective 5: Describe patients that experience severe LFT elevations during lapatanib exposure and calculate the proportion that have lapatanib discontinued and are not re-treated

To achieve these objectives, an observational retrospective cohort study will be conducted using the United States Oncology Electronic Medical Records database. The study population will consist of females with a diagnosis of metastatic breast cancer and a documented order for Lapatanib from January 1, 2007 - December 31, 2009. Patients will be categorized by whether they initiated Lapatanib before or after the July 9, 2008 label change.

'Pre Label': Initiated lapatanib between January 1, 2007 and December 31, 2007. Follow-up time for this group will continue until June 30, 2008 to allow these patients to have at least six months of follow-up time prior to the label change.

'Post Label': Initiated lapatanib between July 9, 2008 and December 31, 2009. Follow-up time for this group will continue until June 30, 2010 to allow these patients to have at least six month of follow-up.

The exposure in this study is lapatanib oral medication. The date of initiation of lapatanib will be the index date. Lapatanib exposure period(s) will be defined from the index date through to the end of the study period (June 30, 2008 for pre-label group or June 30, 2010 for post-label group).

The project will use proportions and two estimates of incidence (cumulative incidence and incidence rates using person-time) to describe the outcomes of interest among the users of Lapatanib before and after the label change. The following LFTs will be considered:

* alanine transaminase (ALT)
* aspartate transaminase (AST)
* alkaline phosphatise (ALP)

ELIGIBILITY:
Inclusion Criteria:

* Female aged >= 19 years
* A diagnosis of breast cancer with documented metastatic disease (as defined by stage at diagnosis, evidence of disease progression, and/or line of therapy);
* Documented order/prescription for lapatanib from January 1, 2007 - December 31, 2009;
* Received care at a practice utilizing the full electronic medical record capabilities of US Oncology's iKnowMed system

Exclusion Criteria:

* Patients participating in clinical trials
* Patients receiving care for another cancer during the study time period

Min Age: 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Female adults age >= 19 years of age with a diagnosis of metastatic breast cancer and who initiated lapatanib from January 1, 2007 - December 31, 2009
Sampling Method: Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2010-12; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
The change in proportion of patients that receive liver function tests prior to the initiation of lapatanib | Within 30 days, 60 days, or 90 days prior to (and including) the day that lapatanib was initiated

SECONDARY OUTCOMES:
The change in prevalence of LFT elevations prior to the initiation of lapatanib | Within 30 days, 60 days or 90 days prior to (and including) the day that lapatanib was initiated
The proportion of patients that have LFT performed routinely (at least every 6 weeks) while exposed to lapatanib | During entire lapatanib exposure (Based on index date between January 2007 - June 2010).
The incidence of LFT elevations while exposed to lapatanib | During entire lapatanib exposure (Based on index date between January 2007 - June 2010).
The proportion of patients with a severe LFT elevation that have lapatanib withdrawn, and are not re-treated | During entire lapatanib exposure (Based on index date between January 2007 - June 2010).

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline